CLINICAL TRIAL: NCT05779644
Title: Effects of GLP-1RA on Body Weight, Metabolism and Fat Distribution in Overweight/Obese Patients With Type 2 Diabetes Mellitus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Jing Ma, Head of Endocrinology and Metabolism, RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT-2022-0245
Record Dates: First submitted 2023-03-09; First posted 2023-03-22 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Metformin; Obesity, Abdominal; Diabetes Mellitus, Type 2; Abdominal Fat; Non-Alcoholic Fatty Liver Disease; Metabolism Disorder, Glucose; Metabolism Disorder, Lipid
Keywords: Metformin; Glucagon-Like Peptide-1 Receptor; Obesity, Abdominal; Diabetes Mellitus, Type 2; Non-Alcoholic Fatty Liver Disease; Metabolism Disorder, Glucose
MeSH Terms: conditions — Obesity, Abdominal; Diabetes Mellitus, Type 2; Non-alcoholic Fatty Liver Disease; Glucose Metabolism Disorders; Lipid Metabolism Disorders | interventions — Liraglutide; semaglutide; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Liraglutide group (Experimental): Liraglutide is injected once a day.
  Interventions: Drug: Liraglutide
- Semaglutide group (Experimental): Semaglutide is injected once a week.
  Interventions: Drug: Semaglutide
- Metformin group (Experimental): Metformin is taken orally daily.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Liraglutide — Liraglutide is injected once a day.
  Arms: Liraglutide group
Drug: Semaglutide — Semaglutide is injected once a week.
  Arms: Semaglutide group
Drug: Metformin — Metformin is taken orally daily.
  Arms: Metformin group

SUMMARY:
The purpose of this study is to analyze the effects of GLP-1RA on blood glucose, body weight, glucose and lipid metabolism and fat distribution in overweight/obese patients with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
Specific research contents: To study the characteristics of glucose and lipid metabolism and fat distribution in overweight/obesity patients with type 2 diabetes mellitus; liraglutide/ semaglutide/ metformin will be applied to patients for one year, and the changes of lipid metabolism and fat distribution in overweight/obese patients with type 2 diabetes and the differences among the three groups will be analyzed before and after treatment. The metabolomic changes of overweight/obese patients with type 2 diabetes before and after medication and the differences among the three groups will be analyzed. Explore the correlation between visceral fat content, glucose and lipid metabolism, inflammatory factors and other biochemical indicators and metabolomics.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65 years old
* BMI≥24kg/㎡, or waist circumference: > 85cm (for male) or > 80cm (for female)
* Has been diagnosed with type 2 diabetes mellitus
* Good blood glucose control in recent three months: random blood sugar < 14mmol/L and HbA1c 6-9%
* Not received any drugs affecting glucose and lipid metabolism or weight loss surgery in the past one month

Exclusion Criteria:

* Abnormal weight gain caused by other endocrine diseases
* Severe metabolic diseases, such as diabetic ketoacidosis, hypertonic hyperglycemia
* Type 1 diabetes or other special types of diabetes
* Used drugs affecting glycolipid metabolism in the past three months
* Severe bleeding tendency that unable to complete venous blood collection
* Patients with MRI contraindications
* Severe renal insufficiency or severe liver insufficiency
* Patients with advanced malignant tumors
* Serious cardiovascular and cerebrovascular diseases
* Rheumatic and immune diseases
* Pregnant and lactating women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-02-23 (Actual); Primary Completion 2025-02-23 (Estimated); Study Completion 2025-02-23 (Estimated)

PRIMARY OUTCOMES:
Blood glucose | The twelfth week of treatment
  Glucose metabolism index
Blood insulin | The twelfth week of treatment
  Glucose metabolism index
Total cholesterol | The twelfth week of treatment
  Lipid metabolism index
Triglyceride | The twelfth week of treatment
  Lipid metabolism index
Lipoprotein | The twelfth week of treatment
  Lipid metabolism index
Weight | The twelfth week of treatment
  Measure fasting weight
Abdominal fat distribution | The twelfth week of treatment
  Use Magnetic resonance imaging-proton density fat fraction to measure fat accumulation in the liver, pancreas and abdomen.

CONTACTS AND LOCATIONS:
Locations (1):
- Ren Ji Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No